CLINICAL TRIAL: NCT04037735
Title: A Clinical Randomized Controlled RSA Trial Comparing the Cemented Attune (S+ Tibia Tray) Fixed Bearing Cruciate Retaining Knee System With the Cemented PFC Sigma Fixed Bearing Cruciate Retaining Knee System
Brief Title: RSA-RCT: Attune S+ TKA Versus Sigma TKA
Acronym: APKnee2-S+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peter den Hollander (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Peter den Hollander, Orthopedic Surgeon, Medical Center Haaglanden
Organization: Medical Center Haaglanden (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P18.131; NL66908.098.18 (Other: https://www.toetsingonline.nl/)
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis Arthritis; Joint Disease; Musculoskeletal Disease; Rheumatic Diseases
Keywords: Comparative Study; Knee Prosthesis; Prosthesis Design; Treatment Outcome; Follow-Up Studies
MeSH Terms: conditions — Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ATTUNE (Experimental): Total Knee Replacement with the ATTUNE S+ Knee Prosthesis by DePuy
  Interventions: Device: ATTUNE S+ Knee Prosthesis by DePuy
- PFC Sigma (Active Comparator): Total Knee Replacement Surgery with PFC Sigma Knee Prosthesis by DePuy
  Interventions: Device: PFC Sigma Knee Prosthesis by DePuy

INTERVENTIONS:
Device: ATTUNE S+ Knee Prosthesis by DePuy — Total Knee Replacement (TKR) Surgery with ATTUNE S+ Knee Prosthesis by DePuy
  Arms: ATTUNE
Device: PFC Sigma Knee Prosthesis by DePuy — Total Knee Replacement Surgery with PFC Sigma Knee Prosthesis by DePuy
  Arms: PFC Sigma

SUMMARY:
The PFC Sigma Knee by DePuy Synthes is an excellent knee replacement with an excellent clinical track record, good survival rates (98% 10 years survival in patients aged < 55 years) and minimal early migration as measured with RSA (0.5mm MTPM at two years follow-up).

The Attune Knee by DePuy Synthes is an advancement in knee replacement options. It is designed to provide better range of motion and address the unstable feeling some patients experience during everyday activities, such as stair descent and bending. To date, more than 470,000 patients have received an Attune Knee and positive feedback was received regarding patient recovery, stability and motion.

The objective of this study is to accurately assess and compare migration, clinical and radiological outcome and patient reported outcomes of two knee prostheses: the Cemented Attune Fixed Bearing Cruciate Retaining Knee System and the Cemented PFC Sigma Fixed Bearing Cruciate Retaining Knee System, both by DePuy Synthes, Warsaw, Indiana, USA. The primary objective of this study is to compare the magnitude and pattern of migration of the prostheses (Femoral and Tibial component). The secondary objective of this study is to compare clinical and radiological outcome of the prostheses and PROMS.

This study is designed as a single-blind, randomized trial between the Attune Knee System and PFC Sigma Knee System. 32 patients with the Attune Knee System and 32 patients with PFC Sigma Knee System will be included in this study.

The study population will consist of patients with symptomatic osteoarthritis of the knee scheduled for knee replacement surgery at the Department of Orthopaedics, Haags Medisch Centrum The Hague (HMC), The Netherlands. Annually 350 TKA procedures are performed in this department, of which about 90% is Osteo Arthritis (OA) and 10% Rheumatoid Arthritis (RA) and other indications. We anticipate that inclusion can be accomplished within a 1 year period and that the total study duration is 3 years.

Main study parameters/endpoints are:

* Migration, measured by means of RSA.
* Patient Reported Outcome Measures by means of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with osteoarthritis and requires primary knee arthroplasty
* All consecutive patients ("usual care") are included to prevent selection bias in the migration analysis.
* Patient is capable of giving informed consent and expressing a willingness to comply with this study

Exclusion Criteria:

* The patient has an a-priori risk for a posterior-stabilized total knee arthroplasty.

  * Insufficiency of the posterior cruciate ligament (PCL)
  * Status after patellectomy
  * In case flexion is less than 90 degrees
  * The patient is diagnosed with Rheumatoid Arthritis
  * When it is expected that the tibia cut during surgery will compromise the attachment of the PCL (because of bony defects)
* The patient is unable or unwilling to sign the Informed Consent specific to this study
* The patient does not understand the Dutch or English language good enough to participate
* Patients indicated for revision arthroplasty instruments because of bone defects or deformity of the bone
* When there are not enough markers visible in the baseline RSA photograph and it will not improve by placing the patient in another position, the patient will be excluded from the study (secondary exclusion criteria).

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Migration, Maximum Total Point Motion (MTPM in mm) measured by means of Radiostereometry (RSA) | 2 Years
  Compare the magnitude and pattern of migration of the prostheses (Tibial and Femoral component, smaller MTPM is better)
  Migration is defined as the relative movement of the prosthesis with respect to the markers in the bone.
  MTPM is defined as Maximum Total Point Motion, which means the amount of motion of the point that moves the most.

SECONDARY OUTCOMES:
EQ-5D with 3 levels of severity for each of the 5 dimensions (EQ-5D-3L) | 2 Years
  General Health: EuroQol 3 Dimensional (EQ-5D) Health Questionnaire measured using patient questionnaire; Index, 0 (worst possible) - 100 (best possible).
Knee injury and Osteoarthritis Outcome Score (KOOS-PS) | 2 Years
  Knee Function: Knee injury and Osteoarthritis Outcome Score (KOOS) measured using patient questionnaire; Index, 0 (worst possible) - 100 (best possible).
Visual Analogue Scale (VAS) pain | 2 Years
  Pain score after activity and during rest; Likert scale 0 (no-pain) -10 (extreme pain).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hollander, MD, Principal Investigator — Haaglanden Medical Center; Rob G Nelissen, Prof., Principal Investigator — Leiden University Medical Center
Locations (1):
- Haaglanden Medical Center, The Hague, South Holland, Netherlands